CLINICAL TRIAL: NCT00005649
Title: An Open-Label Combination Study of Capecitabine and Standard Paclitaxel Therapy as First or Second Line Therapy in Women With Metastatic Breast Carcinoma
Brief Title: Paclitaxel and Capecitabine in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Purpose: Treatment
Other Study IDs: CDR0000067869; ROCHE-M66104C
Record Dates: First submitted 2000-05-02; First posted 2004-04-28 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Paclitaxel

INTERVENTIONS:
Drug: capecitabine
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel and capecitabine in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety, response rate, and efficacy of combination therapy with paclitaxel and capecitabine as first or second line therapy in women with metastatic breast cancer.

OUTLINE: This is a multicenter study. Patients receive paclitaxel IV over 3 hours on day 1 and capecitabine orally twice daily on days 1-14. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed for survival status every 3 months upon completion of treatment.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic breast cancer Bidimensionally measurable disease Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to 75 Sex: Female Menopausal status: Not specified Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: ANC at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) Renal: Creatinine less than 1.5 times ULN Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Eligible patients may have received prior chemotherapy in metastatic or adjuvant setting with the following exceptions: At least 12 months since prior fluoropyrimidine therapy At least 12 months since prior taxane therapy Only 1 previous chemotherapeutic regimen in the metastatic setting Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-07; Primary Completion 2002-07-04 (Actual); Study Completion 2002-07-04

CONTACTS AND LOCATIONS:
Overall Officials: William J. Gradishar, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- PPD Development, Wilmington, North Carolina, United States

REFERENCES:
- [Result] Gradishar WJ, Meza LA, Amin B, Samid D, Hill T, Chen YM, Lower EE, Marcom PK. Capecitabine plus paclitaxel as front-line combination therapy for metastatic breast cancer: a multicenter phase II study. J Clin Oncol. 2004 Jun 15;22(12):2321-7. doi: 10.1200/JCO.2004.12.128. PMID 15197193